CLINICAL TRIAL: NCT05473117
Title: iNav-based, Automated Coronary Magnetic Resonance Angiography for the Detection of Coronary Artery Stenosis (iNav-AUTO CMRA)
Brief Title: iNav-based, Automated Coronary Magnetic Resonance Angiography for the Detection of Coronary Artery Stenosis
Acronym: iNav-AUTO CMRA
Status: Not yet recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Gregory Wood, Dr, University of Aarhus
Other Study IDs: iNav-AUTO CMRA
Record Dates: First submitted 2022-07-19; First posted 2022-07-25 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Coronary Artery Stenosis
Keywords: Coronary Magnetic Resonance Angiography; Coronary Artery Stenosis; Artificial Intelligence
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Group: A single cohort consisting of 230 patients referred for CT Coronary Angiography (CCTA) at risk of coronary artery disease. All patients will undergo both CCTA and CMRA
  Interventions: Diagnostic Test: Coronary Magnetic Resonance Angiography (CMRA)

INTERVENTIONS:
Diagnostic Test: Coronary Magnetic Resonance Angiography (CMRA) — A highly optimised CMRA protocol integrating advanced, automated software for detection of coronary artery stenosis

SUMMARY:
Ischaemic Heart Disease (IHD) is the worlds leading cause of death. IHD is often caused by a narrowing of the coronary arteries, which prevents blood from flowing to the heart muscle, causing pain and damage to the heart. If an individual has a myocardial infarction (MI), parts of the heart that are damaged cannot be repaired. Therefore, it is important to identify and treat the narrowing of the arteries before an MI occurs.

At present there are 2 main methods of identifying narrowing of the arteries. The first is an invasive procedure, the other using a CT scan. Whilst both methods are effective, they entail risk. The invasive procedure can damage the coronary arteries, whilst the CT scan exposes patients to radiation and contrast, which can increase the risk of cancer and allergic reactions.

Magnetic Resonance (MR) scanning is an alternative to these methods, but it has been limited in use in the past due, in part, to the high technical knowledge required to obtain images. In addition, there is a degree of subjectivity in the selection of the mid-diastolic rest period, potentially affecting consistency of results. This means it is difficult to use in a day-to-day hospital environment. However, recent technological developments using artificial intelligence mean that images can be acquired in a more automated and consistent fashion. This new scan has yet to be tested in a clinical trial.

Therefore, the objective of the clinical study is to test this new scan to determine its efficacy. 230 patients at 5 sites at risk of coronary artery disease, who have been referred for invasive coronary angiography, will undergo both their angiography and the new MR scan. The MR scan will then be compared to CCTA for diagnostic accuracy and image quality.

The investigators hypothesise that the new MR scan will have the same diagnostic accuracy as invasive coronary angiography, with no differences in interpretation of the images across the 5 different hospitals.

If proven effective, this would demonstrate that MR scanning of the coronary arteries could prove a safe, clinically useful alternative to both CT scanning and invasive assessment of coronary artery narrowing. In addition, if there is no difference across different locations, it would demonstrate that these scans can be performed consistently, facilitating implementation on a healthcare-system wide basis.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* ≥18 years old
* Subject has provided informed written consent
* BMI < 35
* Sinus Rhythm
* Stable symptom at time of inclusion
* Undergoing CCTA within 28 days

Exclusion Criteria:

* Any contraindication to CMR
* Previous coronary revascularisation
* Inability to take sublingual nitroglycerin
* Irregular heart rate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be drawn from individuals referred to CCTA for assessment of the coronary arteries living in the regions of the 5 study sites, which are based at the following hospitals:
  * Aarhus University Hospital (Aarhus, Denmark)
  * Herlev-Gentofte Hospital (Copenhagen, Denmark)
  * Kings College London (London, UK)
  * Hammersmith Hospital (London, UK)
  * Rigshospitalet (Copenhagen, Denmark)
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Haemodynamically significant CAD | CCTA will take place on clinical indication to investigate risk of CAD following an episode of chest pain. CMRA will be acquired ± 4 weeks compared to CCTA.
  Number of patients with haemodynamically significant CAD, defined as coronary artery diameter stenosis ≥50%, as assessed by CMRA, compared to CCTA.

SECONDARY OUTCOMES:
Image quality | CCTA will take place on clinical indication to investigate risk of CAD following an episode of chest pain. CMRA will be acquired ± 4 weeks compared to CCTA.
  Qualitative assessment of the image quality of the CMRA images. The scale used will be: 0, non-diagnostic; 1, poor (limited coronary vessel visibility or noisy image); 2, average (coronary vessel visible but diagnostic confidence low); 3, good (coronary artery adequately visualised and diagnostic quality image); and 4, excellent (coronary artery clearly depicted).

OTHER OUTCOMES:
Inter-reader variability in interpretation of the CMRA protocol | CCTA will take place on clinical indication to investigate risk of CAD following an episode of chest pain. CMRA will be acquired ± 4 weeks compared to CCTA.
  Number of patients with haemodynamically significant CAD, defined as coronary artery diameter stenosis ≥50%, as assessed by CMRA, as compared between different investigators at different sites in the multi-centre study.
Pulse rate | CCTA will take place on clinical indication to investigate risk of CAD following an episode of chest pain. CMRA will be acquired ± 4 weeks compared to CCTA.
  Pulse during CMRA scan acquisition and association with image quality metrics

CONTACTS AND LOCATIONS:
Overall Officials: Won Yong Kim, Study Chair — Department of Cardiology, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Wood G, Hajhosseiny R, Pedersen AU, Littlewood S, Hansen TJ, Neji R, Kunze KP, Wetzl J, Norgaard BL, Jensen JM, Maeng M, Madsen PL, Vejlstrup N, Prieto C, Botnar RM, Kim WY. Image navigator-based, automated coronary magnetic resonance angiography for the detection of coronary artery stenosis. J Cardiovasc Magn Reson. 2024 Winter;26(2):101097. doi: 10.1016/j.jocmr.2024.101097. Epub 2024 Sep 16. PMID 39293786